CLINICAL TRIAL: NCT05359731
Title: Pharmacokinetic Analysis of Bupivacaine in the Presence and Absence of Perineural Dexamethasone in Axillary Brachial Plexus Blockade for Distal Forearm and Hand Surgery
Brief Title: Pharmacokinetic Analysis of Bupivacaine in the Presence and Absence of Perineural Dexamethasone in Axillary Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Daniela Bravo Advis, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OAIC 1249/22
Record Dates: First submitted 2022-04-28; First posted 2022-05-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Analgesia; Acute Pain; Upper Extremity Injury
Keywords: Dexamethasone; Nerve Block; Adjuvant; Pharmacokinetic Analysis
MeSH Terms: conditions — Agnosia; Acute Pain; Arm Injuries | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A research assistant (licensed anesthesiologist) will prepare the local anesthetic solutions and will add the study drug following the randomization order. The operator, patient and investigator assessing the block will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineural Bupivacaine (Active Comparator): Bupivacaine without Dexamethasone in axillary brachial plexus blockade
  Interventions: Drug: Bupivacaine Hydrochloride
- Perineural Bupivacaine plus Dexamethasone (Experimental): Bupivacaine with Dexamethasone in axillary brachial plexus blockade
  Interventions: Drug: Bupivacaine Hydrochloride with Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Patients will receive a total volume of 30 ml of bupivacaine 0.5% in an axillary block with a double puncture.
  Arms: Perineural Bupivacaine
Drug: Bupivacaine Hydrochloride with Dexamethasone — Patients will receive a total volume of 30 ml of bupivacaine 0.5% with Dexamethasone 4 mg in an axillary block with a double puncture.
  Arms: Perineural Bupivacaine plus Dexamethasone

SUMMARY:
The investigators will conduct a prospective, randomized, double-blinded study using an axillary brachial plexus block in patients undergoing elective surgery of the distal forearm and hand to characterize and describe the pharmacokinetics of bupivacaine associated with perineural dexamethasone.

The pharmacokinetic analysis will be performed by measuring bupivacaine plasma levels at different time intervals after the blockade (15, 30, 45, 60, and 90 minutes), allowing comparison between 2 different groups: Bupivacaine (B) and Bupivacaine-dexamethasone (BD).

Thus, the hypothesis is that plasma levels of bupivacaine during the first 90 minutes after a blockade are lower in the presence of perineural dexamethasone, suggesting a decrease, at least initially, in systemic absorption from the injection site.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification 1-2
* Real weight between 80 and 100 kg
* Body mass index between 20 and 30

Exclusion Criteria:

* Adults who are not capable of giving their own consent
* Medical history or physical findings of pre-existing neuropathy
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs)
* Pregnancy
* Previous surgery in the axillary region of the surgical side

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of bupivacaine | 0 to 90 minutes after the ending time of local anesthetic injection
  Maximum plasmatic level of bupivacaine

SECONDARY OUTCOMES:
Plasmatic concentration of bupivacaine at 15 minutes | 15 minutes after the ending time of local anesthetic injection
  Plasmatic level of bupivacaine 15 minutes after local anesthetic injection (ng/ml)
Plasmatic concentration of bupivacaine at 30 minutes | 30 minutes after the ending time of local anesthetic injection
  Plasmatic level of bupivacaine 30 minutes after local anesthetic injection (ng/ml)
Plasmatic concentration of bupivacaine at 45 minutes | 45 minutes after the ending time of local anesthetic injection
  Plasmatic level of bupivacaine 45 minutes after local anesthetic injection (ng/ml)
Plasmatic concentration of bupivacaine at 60 minutes | 60 minutes after the ending time of local anesthetic injection
  Plasmatic level of bupivacaine 60 minutes after local anesthetic injection (ng/ml)
Plasmatic concentration of bupivacaine at 90 minutes | 90 minutes after the ending time of local anesthetic injection
  Plasmatic level of bupivacaine 90 minutes after local anesthetic injection (ng/ml)
Time to obtain the maximum plasma concentration of bupivacaine (Tmax) | 0 to 90 minutes after the ending time of local anesthetic injection
  Time in minutes in which the maximum plasmatic level of bupivacaine is reached
Area under the curve of plasma concentration versus time at 90 minutes (AUC90) | 0 to 90 minutes after the ending time of local anesthetic injection
  Area under the curve at 90 minutes
Sensory and motor block score | 30 minutes after the ending time of local anesthetic injection
  The sensorimotor block will be assessed every 5 minutes until 30 minutes after the end of local anesthetic injection using a 16-point composite score evaluating sensory and motor block of musculocutaneous, medium, radial, and ulnar nerves.
  Sensation will be assessed with ice in each nerve territory with a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, the patient can feel touch but not cold; 2= anesthetic block, the patient cannot feel cold or touch.
  The motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
  Successful blocks at 30 minutes correlate with a final score ( sum of all individual sensory and motor scores) of at least 14 points out of 16.
Block onset time | 30 minutes after the ending time of local anesthetic injection
  Time required to reach a minimal sensorimotor composite score of 14 points out of a maximum of 16 points. The sensorimotor score is described in outcome 9.
Incidence of successful block | 30 minutes after the ending time of local anesthetic injection
  Percentage of blocks with a minimal sensorimotor composite score of 14 points out of a maximum of 16 points at 30 minutes after the injection
Motor block duration | 48 hours after the ending time of local anesthetic injection
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of return of hand and fingers movement.
Sensory block duration | 48 hours after the ending time of local anesthetic injection
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of the return of hand and fingers sensation
Analgesic block duration | 48 hours after the ending time of local anesthetic injection
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of the first sensation of pain in the surgical area
Intensity of pain during block procedure | During the execution of the nerve blockade
  Evaluated with the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-points score represents the worst imaginable pain. Patients will be asked to rate their pain verbally with this scale. The blinded assessor will register the score reported.
Block performance time | From the skin anesthesia to the end of local anesthetic injection
  Sum of: 1- the acquisition time of the ultrasonographic image. and 2- the time to perform the block itself (from the skin anesthesia to the end of local anesthetic injection)
Incidence of nerve block side effects | From the skin anesthesia to the end of local anesthetic injection
  Determined by the presence of paresthesia, local anesthetic systemic toxicity, vascular puncture after the block.
Persistent neurologic deficit | 7 days after surgery
  Presence of persistent sensory or motor postoperative deficit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Metropolitan, Chile

REFERENCES:
- [Background] Desai N, Albrecht E, El-Boghdadly K. Perineural adjuncts for peripheral nerve block. BJA Educ. 2019 Sep;19(9):276-282. doi: 10.1016/j.bjae.2019.05.001. Epub 2019 Jul 6. No abstract available. PMID 33456903
- [Background] Leurcharusmee P, Aliste J, Van Zundert TC, Engsusophon P, Arnuntasupakul V, Tiyaprasertkul W, Tangjitbampenbun A, Ah-Kye S, Finlayson RJ, Tran DQ. A Multicenter Randomized Comparison Between Intravenous and Perineural Dexamethasone for Ultrasound-Guided Infraclavicular Block. Reg Anesth Pain Med. 2016 May-Jun;41(3):328-33. doi: 10.1097/AAP.0000000000000386. PMID 27015546
- [Background] Aliste J, Leurcharusmee P, Engsusophon P, Gordon A, Michelagnoli G, Sriparkdee C, Tiyaprasertkul W, Tran DQ, Van Zundert TC, Finlayson RJ, Tran DQH. A randomized comparison between intravenous and perineural dexamethasone for ultrasound-guided axillary block. Can J Anaesth. 2017 Jan;64(1):29-36. doi: 10.1007/s12630-016-0741-8. Epub 2016 Sep 23. PMID 27663451
- [Background] Heesen M, Klimek M, Imberger G, Hoeks SE, Rossaint R, Straube S. Co-administration of dexamethasone with peripheral nerve block: intravenous vs perineural application: systematic review, meta-analysis, meta-regression and trial-sequential analysis. Br J Anaesth. 2018 Feb;120(2):212-227. doi: 10.1016/j.bja.2017.11.062. Epub 2017 Nov 22. PMID 29406171
- [Background] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271
- [Background] Shishido H, Kikuchi S, Heckman H, Myers RR. Dexamethasone decreases blood flow in normal nerves and dorsal root ganglia. Spine (Phila Pa 1976). 2002 Mar 15;27(6):581-6. doi: 10.1097/00007632-200203150-00005. PMID 11884905
- [Background] Gonzalez AP, Bernucci F, Pham K, Correa JA, Finlayson RJ, Tran DQ. Minimum effective volume of lidocaine for double-injection ultrasound-guided axillary block. Reg Anesth Pain Med. 2013 Jan-Feb;38(1):16-20. doi: 10.1097/AAP.0b013e3182707176. PMID 23146999
- [Background] Kirkham KR, Jacot-Guillarmod A, Albrecht E. Optimal Dose of Perineural Dexamethasone to Prolong Analgesia After Brachial Plexus Blockade: A Systematic Review and Meta-analysis. Anesth Analg. 2018 Jan;126(1):270-279. doi: 10.1213/ANE.0000000000002488. PMID 28922230
- [Background] Souza MCO, Marques MP, Duarte G, Lanchote VL. Analysis of bupivacaine enantiomers in plasma as total and unbound concentrations using LC-MS/MS: Application in a pharmacokinetic study of a parturient with placental transfer. J Pharm Biomed Anal. 2019 Feb 5;164:268-275. doi: 10.1016/j.jpba.2018.10.040. Epub 2018 Oct 23. PMID 30399533
- [Background] Tran DQ, Dugani S, Dyachenko A, Correa JA, Finlayson RJ. Minimum effective volume of lidocaine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):190-4. doi: 10.1097/AAP.0b013e31820d4266. PMID 21270721
- [Background] Bravo D, Aliste J, Layera S, Fernandez D, Leurcharusmee P, Samerchua A, Tangjitbampenbun A, Watanitanon A, Arnuntasupakul V, Tunprasit C, Gordon A, Finlayson RJ, Tran DQ. A multicenter, randomized comparison between 2, 5, and 8 mg of perineural dexamethasone for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2019 Jan;44(1):46-51. doi: 10.1136/rapm-2018-000032. PMID 30640652
- [Background] Ferraro LHC, Takeda A, Barreto CN, Faria B, Assuncao NA. [Pharmacokinetic and clinical effects of two bupivacaine concentrations on axillary brachial plexus block]. Braz J Anesthesiol. 2018 Mar-Apr;68(2):115-121. doi: 10.1016/j.bjan.2017.09.001. Epub 2017 Oct 16. PMID 29042063
- [Derived] Bravo D, Aguilera G, Giordano A, Layera S, Erpel H, Mora D, Ramirez C, Jara A, Aliste J. Bupivacaine pharmacokinetics in the absence or presence of perineural dexamethasone in axillary blockade. Br J Anaesth. 2026 Jan 16:S0007-0912(25)00894-3. doi: 10.1016/j.bja.2025.12.009. Online ahead of print. PMID 41547610